CLINICAL TRIAL: NCT02729155
Title: Efficacy of Single-cycle Remote Ischemic Pre/Post-conditioning, for Prevention of Contrast-induced Acute Kidney Injury in Patients With Chronic Kidney Disease Undergoing Coronary Angiography or Coronary Angioplasty
Brief Title: Single-cycle Remote Ischemic Preconditioning and Postconditioning for Prevention of Contrast-Induced Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Principal Investigator, Col. Suthee Panichkul, Phramongkutklao College of Medicine and Hospital, Phramongkutklao College of Medicine and Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: PMK-SCRIP-CIN
Record Dates: First submitted 2016-03-31; First posted 2016-04-06 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Ischemic Reperfusion Injury
Keywords: Ischemic Preconditioning; Postconditioning; Angioplasty; Angiography; Contrast-Induced Nephropathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- RIPre + RIPost (Experimental): Intervention: RIPre 200 mmHg + RIPost 200 mmHg
  Interventions: Procedure: RIPre; Procedure: RIPost
- RIPre + Sham (Experimental): Intervention: RIPre 200 mmHg + Sham 10 mmHg
  Interventions: Procedure: RIPre; Procedure: Sham-Post
- Sham + RIPost (Experimental): Intervention: Sham 10 mmHg + RIPost 200 mmHg
  Interventions: Procedure: RIPost; Procedure: Sham-Pre
- Sham + Sham (Sham Comparator): Intervention: Sham 10 mmHg + Sham 10 mmHg
  Interventions: Procedure: Sham-Pre; Procedure: Sham-Post

INTERVENTIONS:
Procedure: RIPre — Preconditioning 200 mmHg x 5 minutes before procedure
  Arms: RIPre + RIPost; RIPre + Sham
Procedure: RIPost — Postconditioning 200 mmHg x 5 minutes after procedure
  Arms: RIPre + RIPost; Sham + RIPost
Procedure: Sham-Pre — Sham 10 mmHg x 5 minutes before procedure
  Arms: Sham + RIPost; Sham + Sham
Procedure: Sham-Post — Sham 10 mmHg x 5 minutes after procedure
  Arms: RIPre + Sham; Sham + Sham

SUMMARY:
This trial is a 2 x 2 factorial design, double-blinded, randomized controlled trial to evaluate efficacy and safety of remote ischemic preconditioning and postconditioning for prevention of contrast-induced acute kidney injury in patient undergoing coronary angiography and angioplasty

DETAILED DESCRIPTION:
randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* The patient have indication for coronary angiography or angioplasty.
* Impaired renal function with reduced eGFR < 60 ml/min/1.73 m2 by CKD-EPI equation.
* Written informed consent.

Exclusion Criteria:

* History of contrast allergy.
* The patient had end-stage renal failure with the need for hemodialysis.
* The patient take medications that affect the kidneys function within 48 hours before study.
* The patient had acute kidney injury from any cause.
* The patient was received contrast media within 2 weeks before study.
* The patient had cardiac arrest or shock.
* The patient had peripheral arterial disease (PAD)
* Pregnancy
* Refused to study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 596 (Estimated)
Dates: Start 2015-10; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of CI-AKI, which was defined as an increment of serum creatinine 0.5 mg/dL or a relative increase of 25% over the baseline value | Within a period of 24 hours after contrast medium administration

SECONDARY OUTCOMES:
Change in sCr and eGFR from baseline | Within a period of 24 hours after contrast medium administration
Major adverse cerebrovascular and cardiovascular events (MACCE) in each intervention group | Within a period of 6 months after contrast medium administration
  MACCE were composite of death, hospitalization, acute coronary syndrome, congestive heart failure and stroke or transient ischemic attack
Incidence(%) of CI-AKI in differrent subgroups of patient characteristics | Within a period of 24 hours after contrast medium administration
  Patient characteristics include eGFR, global CIAKI risk score, contrast media volume and DM.
  Incidence of CI-AKI, which was defined as an increment of serum creatinine 0.5 mg/dL or a relative increase of 25% over the baseline value.
Incidence(%) of CI-AKI in patients with vs without RIPre and RIPost | Within a period of 24 hours after contrast medium administration
  Incidence of CI-AKI, which was defined as an increment of serum creatinine 0.5 mg/dL or a relative increase of 25% over the baseline value
Incidence(%) of MACCE in differrent subgroups of patient characteristics | Within a period of 6 months after contrast medium administration
  Patient characteristics include eGFR, global CIAKI risk score, contrast media volume and DM.
  MACCE were composite of death, hospitalization, acute coronary syndrome, congestive heart failure and stroke or transient ischemic attack
Incidence(%) of MACCE in patients with vs without RIPre and RIPost | Within a period of 6 months after contrast medium administration
  Patient characteristics include eGFR, global CIAKI risk score, contrast media volume and DM.
  MACCE were composite of death, hospitalization, acute coronary syndrome, congestive heart failure and stroke or transient ischemic attack
Incidence(%) of MACCE in patients who have CI-AKI vs patients who have no CI-AKI | Within a period of 6 months after contrast medium administration
  Incidence of CI-AKI, which was defined as an increment of serum creatinine 0.5 mg/dL or a relative increase of 25% over the baseline value within a period of 24 hours after contrast medium administration

CONTACTS AND LOCATIONS:
Overall Officials: Nakarin Sansanayudh, MD,PhD, Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (1):
- Department of Internal Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes